CLINICAL TRIAL: NCT01759823
Title: Efficacy and Safety of Autologous Bone Marrow Derived Stem Cell Transplantation in Patients With Type 2 Diabetes Mellitus
Brief Title: Bone Marrow Derived Stem Cell Transplantation in T2DM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, Professor and HOD, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: stem cell therapy in T2DM
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- mesenchymal stem cell transplantation (Experimental): Patients with Type 2 Diabetes mellitus on full doses of Vildagliptin+Pioglitazone+Metformin and requiring Insulin at dose of >0.4unit/Kg for blood glucose control.
  Interventions: Biological: mesenchymal stem cell transplantation
- Control (Sham Comparator): vildagliptin+metformin+pioglitazone and on Insulin >0.4unit/Kg who will act as active control.They will receive injectable placebo at Day 1 in addition to above and will be followed up for 6 months.Follow up investigation and Insulin dose titration will be similar to Group 1
  Interventions: Other: control
- MNC's TRANSPLANTATION (Experimental): Patients with Type 2 Diabetes mellitus on full doses of Vildagliptin+Pioglitazone+Metformin and requiring Insulin at dose of >0.4unit/Kg for blood glucose control.
  Interventions: Biological: MNC's TRANSPLANTATION

INTERVENTIONS:
Biological: mesenchymal stem cell transplantation — 20 - 30 ml of bone marrow will be aspirated and layered on density gradient medium (Ficoll - hypaque ) and stem cells will be separated. Separated mono nucleated cells will be dissolved in minimum essential medium and inoculated in culturing flask and mesenchymal will be allowed to adhere to culturing flask and mesenchymal stem cell will be injected into superior pancreatic duodenal artery . Patients will be urged to monitor and document blood glucose readings for next 6 months. Glucagon stimulated C - peptide HYPERGLYCEMIC CLAMP FOR ASSESSMENT OF BETA CELL FUNCTION , Homeostasis Model of Assessment - Insulin Resistance and Beta cell function ,HbA1c, lipid profile and biochemistry will be done at baseline and 6 months .
  Arms: mesenchymal stem cell transplantation
Other: control — 5 ml of bone marrow will be aspirated and 3 mL of Vitamin B complex will be injected through transfemoral route into superior pancreatico-duodenal artery. Patients will be urged to monitor and document blood glucose readings for next 6 months. Glucagon stimulated C - peptide,HYPERGLYCEMIC CLAMP TO ASSESS BETA CELL FUNCTION. Homeostasis Model of Assessment - Insulin Resistance and Beta cell function ,HbA1c, lipid profile and biochemistry will be done at baseline and 6 months .
  Arms: Control
Biological: MNC's TRANSPLANTATION — 20 - 30 ml of bone marrow will be aspirated and layered on density gradient medium (Ficoll - hypaque ) and stem cells will be separated. Separated mono nucleated cells will injected into superior pancreatico duodenal artery. Patients will be urged to monitor and document blood glucose readings for next 6 months. Glucagon stimulated C - peptide HYPERGLYCEMIC CLAMP FOR ASSESSMENT OF BETA CELL FUNCTION , AND EUGLYCEMIC CLAMP TO ASSESS INSULIN SENSITIVITY .Homeostasis Model of Assessment - Insulin Resistance and Beta cell function ,HbA1c, lipid profile and biochemistry will be done at baseline and 6 months .
  Arms: MNC's TRANSPLANTATION

SUMMARY:
The purpose of this study is to improve the blood glucose level in type 2 diabetic patients.

DETAILED DESCRIPTION:
We hypothesize that Autologous bone marrow derived stem cells which would be expanded into culture and their subsequent transplant into the pancreas of patients with T2DM, aged 30 - 70 years with triple oral hypoglycemic agent failure and on insulin(>0.4 U/ kg body weight/day) will lead to abolition or reduction of insulin requirement by more than or equal to 50% in these patients over a period of 6 months. It is assumed that stem cell in these patients leads to increased angiogenesis, secretion of various cytokines and upregulation of pancreatic transcription factors and Vascular endothelial growth factor(VEGF) and creates a micro-environment which supports beta cell/resident stem cell activation and survival.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes mellitus between 30 and 70 years of age.

* Failure to triple oral hypoglycemic agent and on stable doses of insulin for at least 3 months.
* On vildagliptin,pioglitazone and metformin for at least 3 months along with Insulin to maintain euglycemia.
* HbA1c < 7.5%.
* Insulin requirement ≥0.4 IU/kg/d.
* GAD antibody negative status.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus or secondary diabetes.
* Patients with serum creatinine > 1.5 mg/dl.
* Abnormal liver function tests (defined as value of transaminases > 3 times the upper value of normal or serum bilirubin higher than normal for the reference value for the laboratory).
* History of cholecystitis/ cholelithiasis/ cholecystectomy
* Seropositivity for HIV, HBsAg and hepatitis C virus (HCV).
* History of myocardial infarction or unstable angina in the previous 3 months.
* History of malignancy
* Patients with active infections.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Reduction of insulin requirement by ≥ 50% by the end of 6 months of autologous bone marrow derived stem cell transplantation and Improvement in Glucagon stimulated C - peptide levels and hyperglycemic clamp for assessment of beta cell function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: A Bhansali, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; V Jha, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Neelam Marwaha, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Uttarakhand, India

REFERENCES:
- [Background] Bhansali A, Upreti V, Khandelwal N, Marwaha N, Gupta V, Sachdeva N, Sharma RR, Saluja K, Dutta P, Walia R, Minz R, Bhadada S, Das S, Ramakrishnan S. Efficacy of autologous bone marrow-derived stem cell transplantation in patients with type 2 diabetes mellitus. Stem Cells Dev. 2009 Dec;18(10):1407-16. doi: 10.1089/scd.2009.0164. PMID 19686048
- [Derived] Bhansali S, Dutta P, Yadav MK, Jain A, Mudaliar S, Hawkins M, Kurpad AV, Pahwa D, Yadav AK, Sharma RR, Jha V, Marwaha N, Bhansali S, Bhansali A. Autologous bone marrow-derived mononuclear cells transplantation in type 2 diabetes mellitus: effect on beta-cell function and insulin sensitivity. Diabetol Metab Syndr. 2017 Jul 4;9:50. doi: 10.1186/s13098-017-0248-7. eCollection 2017. PMID 28690682